CLINICAL TRIAL: NCT00540787
Title: A Randomized Comparison of the Efficacy of Antiarrhythmic Drug Therapy and Radiofrequency Catheter Ablation for the Maintenance of Sinus Rhythm In Patients With Paroxysmal Atrial Fibrillation
Brief Title: A Comparison of Antiarrhythmic Drug Therapy and Radio Frequency Catheter Ablation in Patients With Paroxysmal Atrial Fibrillation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: A4
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation; Amiodarone; Flecainide; Propafenone; Quinidine; dofetilide; Sotalol; cifenline; Calcium Channel Blockers; Anti-Arrhythmia Agents

ARMS (2):
- Drug Treatment (Active Comparator)
  Interventions: Device: Radiofrequency ablation, antiarrhythmic drugs; Drug: Amiodarone, flecainide, propafenone, quinidine, dofetilide, sotalol, cibenzoline, beta blocking and calcium channel blocking agents and antiarrhythmic drugs
- ThermoCool Radiofrequency Catheter (Active Comparator): Radiofrequency catheter used.
  Interventions: Device: Radiofrequency ablation, antiarrhythmic drugs; Device: ThermoCool Radiofrequency Catheter

INTERVENTIONS:
Device: Radiofrequency ablation, antiarrhythmic drugs — Patients receive either treatment.
Drug: Amiodarone, flecainide, propafenone, quinidine, dofetilide, sotalol, cibenzoline, beta blocking and calcium channel blocking agents and antiarrhythmic drugs — Amiodarone will be taken at 600 mg per day for 21 days (as a loading dose) followed by 1.4g per week or 200mg per day. The daily dose may be increased to 300mg or 2.1g per week.
  Arms: Drug Treatment
Device: ThermoCool Radiofrequency Catheter — Patient is ablated once, repeat ablation if paroxysmal atrial fibrillation reoccurs.
  Arms: ThermoCool Radiofrequency Catheter

SUMMARY:
The purpose of this study is to compare radiofrequency catheter ablation and antiarrhythmic drug treatment for the maintenance of sinus rhythm in paroxysmal atrial fibrillation patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Paroxysmal atrial fibrillation for at least 6 months with at least 2 symptomatic episodes (patient history) during the previous month
* Atrial fibrillation (patient history or echocardiogram documented) resistant to at least one antiarrhythmic drug of Class I or III
* Documentation of at least one episode of atrial fibrillation on 12-lead echocardiogram or Holter Monitor

Exclusion Criteria:

* Contraindications to more than 2 antiarrhythmic drugs of different classes, or to oral anticoagulants
* History of any previous ablation for atrial fibrillation
* Intracardiac thrombus
* Atrial fibrillation due to reversible cause
* Pregnancy
* Contraindication to stopping oral anticoagulation (for example as a result of a mechanical cardiac valve)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2003-08-01 (Actual); Primary Completion 2006-06-01 (Actual); Study Completion 2006-06-01 (Actual)

PRIMARY OUTCOMES:
Recurrence of Atrial Fibrillation | One year
  To compare the incidence of recurrence of Atrial Fibrillation in the two groups over a follow-up period of one year.

SECONDARY OUTCOMES:
Efficacy of ablation and drug treatment | One year
  Evaluation of:
  * the functional state of the 2 groups of patients in terms of quality of life
  * the efficacy of the subgroup receiving amiodarone as compared to curative ablation
  * the incidence of secondary effects of both approaches
  * the rate of withdrawal from oral anticoagulation at 1 year after randomization
  * the effect of ablation for maintenance of sinus rhythm with previously ineffective drugs in case of failure of ablation strategy (after cross-over to medical treatment)
  * the assessment of Atrial fibrillation burden in both groups (using patient diaries and Holter Monitors)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Jais, MD, Principal Investigator — Hôpital Haut Lèvêque
Locations (6):
- United States (3):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mid-Ohio Cardiology, Columbus, Ohio
- France (2):
  - Hôpital Haut Lèvêque, Pessac, Paris
  - Hopital Lariboisiere, Paris
- Hopital Cantonal de Geneve, Geneva, Switzerland

REFERENCES:
- [Derived] Jais P, Cauchemez B, Macle L, Daoud E, Khairy P, Subbiah R, Hocini M, Extramiana F, Sacher F, Bordachar P, Klein G, Weerasooriya R, Clementy J, Haissaguerre M. Catheter ablation versus antiarrhythmic drugs for atrial fibrillation: the A4 study. Circulation. 2008 Dec 9;118(24):2498-505. doi: 10.1161/CIRCULATIONAHA.108.772582. Epub 2008 Nov 24. PMID 19029470